CLINICAL TRIAL: NCT01828580
Title: Safety and Performance Evaluation of the AutoLap System - a Feasibility Study
Brief Title: Safety and Performance Evaluation of the AutoLap System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.S.T. Medical Surgery Technology LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AL-65-001
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Patients Scheduled for Hernia Repair, Cholecystectomy, Right Colectomy, Nissen Fundoplication and Sigmoid Resection
Keywords: laparoscopic Cholecystectomy; Gallbladder removal; laparoscope holder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AutoLap (Experimental)
  Interventions: Device: active laparoscope positioner (AutoLap)

INTERVENTIONS:
Device: active laparoscope positioner (AutoLap)

SUMMARY:
The main objectives of this study are to evaluate the safety and performance of the AutoLap system in Laparoscopic Cholecystectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form.
2. Patients between 18 and 75 years of age inclusive who were scheduled for elective laparoscopic Cholecystectomy procedure.

Exclusion Criteria:

1. Previous upper abdominal surgery and contraindications to Pneumoperitoneum.
2. Pregnancy.
3. Obesity (BMI >35 Kg/m2).
4. Generalized peritonitis.
5. Septic shock from cholangitis.
6. Severe acute pancreatitis.
7. Uncorrected coagulopathy.
8. Previous abdominal operations which prevent safe abdominal access or progression of the procedure.
9. Advanced cirrhosis with failure of hepatic function.
10. Suspected gallbladder cancer.
11. Acute cholecystitis
12. Presence of any medical or psychiatric condition or any other condition that, in the opinion of the Investigator, could affect the successful participation of the patient in the study.
13. Patient participates in any other clinical study 60 days prior to the start of the study and throughout the study duration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | participants will be followed for the duration of hospital stay, an expected average of 1-2 days
  No conversion to open surgery from laparoscopic surgery due to using the AutoLap system 2) No AutoLap system related operative complications, that require further clinical intervention
Performance evaluation | during surgery -defined as the time from the first abdominal incision until the surgical procedure is completed (skin incisions are closed).
  The ability of the AutoLap system to successfully move the laparoscope to the surgeon's desired position

SECONDARY OUTCOMES:
system set-up time | during surgery - defined as the time from the first abdominal incision until the surgical procedure is completed (skin incisions are closed).
  defined as the time required from connecting the AutoLap's ARM to the bed rail
Average total procedure time | during surgery - defined as the time from the first abdominal incision until the surgical procedure is completed (skin incisions are closed).
  defined as the time from first abdominal incision until the surgical procedure is completed
Number of times that the laparoscope was removed for cleaning | During surgery - defined as the time from the first abdominal incision until the surgical procedure is completed (skin incisions are closed).
Usability evaluation | During surgery (at the end of the procedure)
  the AutoLap system usability in laparoscopic procedures will be assessed by a questionnaire. The questionnaire assesses the surgeon's satisfaction with the use of the AutoLap in regard to easiness of use, convenient of movement control and its ability to be used in the OR without interfering with the surgical flow

CONTACTS AND LOCATIONS:
Locations (3):
- Assuta Medical Center, Tel Aviv, Israel, Israel
- Niguarda Cà Granda Hospital, Milan, Italy
- Meander Medisch Centrum, Amersfoort, Netherlands